CLINICAL TRIAL: NCT03596125
Title: Correction of Neonatal Glutathione by N-acetylcysteine in Pregnant Women at Risk of Premature Birth
Brief Title: Correction of Neonatal Glutathione by N-acetylcysteine in Pregnant Women at Risk of Premature Birth (GSH MAP)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: difficulty of recruitment
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC15_0476
Record Dates: First submitted 2018-05-28; First posted 2018-07-23 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Preterm Delivery
Keywords: Glutathione; Antioxidant; Oxidative stress; Preterm
MeSH Terms: conditions — Premature Birth | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine (NAC) (Experimental): High risk of prematurity: 9g intravenously then 6g (per os) a day until day 7, then 1,8g (per os) a day until 37 weeks of gestational age.
  Moderate risk of prematurity: 6g (per os) a day until day 7 then 1,8g ( per os) a day until 37 weeks of gestational age.
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): High risk of prematurity: 9g intravenously then 6g (per os) a day until day 7, then 1,8g (per os) a day until 37 weeks of gestational age.
  Moderate risk of prematurity: 6g (per os) a day until day 7 then 1,8g ( per os) a day until 37 weeks of gestational age.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine supplementation
  Other Names: NAC
  Arms: N-acetylcysteine (NAC)
Drug: Placebo — per os: jelly tablets Intravenous Route: Glucidion G5
  Arms: Placebo

SUMMARY:
Birth exposes the newborn to oxidative stress, as due to the switch from a protected, relatively hypoxic intrauterine milieu into an environment with a high oxygen pressure. The full-term newborn is well prepared to this massive redox challenge at the time of birth due to his well-integrated antioxidant defenses. On the contrary, numerous bibliographical data and our own work demonstrate the fragility of preterm newborns in this context of oxidative stress, linked to the immaturity of his antioxidant defenses.

Premature birth abruptly propels the fetus from the protected, relatively hypoxic intrauterine milieu to an environment at risk of free radical injury caused by mechanical ventilation strategies, including the use of high inspired oxygen fractions or inhaled nitric oxide, generating excessive reactive oxidative species (ROS). Several studies highlight the key role of ROS in adverse outcomes of preterm infant suffering from low birth weight, bronchopulmonary dysplasia, necrotizing enterocolitis or retinopathy.

This project aims to evaluate a therapeutic anti-oxidative strategy in order to correct the oxidative status of preterm infants. The investigators propose an early intervention that consists in an antenatal maternal supplementation with N-acetylcysteine (NAC), the acetylated precursor of both cysteine and glutathione, a key physiological antioxidant. This strategy could be promising for the development of simplified and personalized care of preterm infants.

GSH MAP is a randomized, single-blind, placebo-controlled study that aims to determine if NAC supplementation in women admitted to hospital care due to preterm labor (prior to 34 weeks of gestational age) may correct glutathione deficiency in neonatal cord blood.

DETAILED DESCRIPTION:
GSH MAP is a randomized single-blind, placebo-controlled study. The design will include the recruitment of 120 pregnant women admitted to hospital care due to preterm labor (above 18 yrs of age, gestational age between 24 and 34 weeks). According to the risk of preterm delivery, women will be treated following two different schedules :

* High risk of prematurity: NAC supplementation -9 g intravenously-6g/day per os until day 7-1,8g/day per os until 37 weeks of gestational age.
* Moderate risk of prematurity: NAC supplementation -6g/day per os until day 7-1,8g/day per os until 37 weeks of gestational age.

Biological samples collected: maternal blood at inclusion, maternal/cord blood and placenta at delivery, breast milk samples during the first week of lactation in case of exclusive breastfeeding.

Levels of glutathione and related metabolites will be measured in plasma, red blood cells, placenta and breast milk.

In ancillary studies, metabolome and lipidome profilings will be performed on maternal and cord blood and on breast milk samples.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Moderate or severe risk of prematurity
* Mono-fetal pregnancy
* And a term of pregnancy > = 24 weeks and <34 weeks of gestation at diagnosis
* subjects affiliated with an appropriate social security system
* written signed informed consent form

Exclusion Criteria:

* Age < 18 years old
* Major under trusteeship or curatorship
* Maternal refusal and / or Incapacity to understand the benefits and potential risks of the protocol and to sign an informed consent form.
* A sonographic cervix ≥ 20 mm
* Mothers WITH:

  * A Body mass index less than 18 kg/m2 and greater than 40 kg/m2 before pregnancy
  * Type I, II diabetes
  * Epileptic disorders
  * A history of asthma
  * A hemorrhagic pathology
  * Maternal infection (HIV, hepatitis B and C) other than chorioamnionitis
* Patients in labour treated with magnesium sulphate
* Multiple pregnancy
* A known allergy/ hypersensitivity to N-acetylcysteine
* Fetal pathology other than intrauterine growth retardation (such as: karyotype abnormality, malformation, intrauterine growth retardation <10th percentile)
* Current high doses of antioxidants treatments (vitamin supplements, ...)
* Patient with proven pre-eclampsia
* Patient with heart failure
* Patient with nephropathy
* Patient with medically known lactose intolerance
* Patient not affiliated with an appropriate social security system

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Venous umbilical cord blood concentration of glutathione (micromoles/L) following antenatal NAC supplementation. | 13 weeks
  The venous umbilical cord blood concentration of glutathione will be measured in red blood cell lysates on C18-reverse phase column using liquid-chromatography combined to mass spectrometry. Homocysteine, cysteine, reduced (GSH) and oxidized (GSSG) glutathione levels will be measured in erythrocytes by comparing an experimental arm versus a placebo arm

SECONDARY OUTCOMES:
Number of days between the NAC-therapeutic initialization and childbirth. | until childbirth
  The delay time (days) between delivery and inclusion of pregnant women admitted to hospital care due to preterm labor will be compared in an experimental arm versus a placebo arm.
Glutathione concentration in arterial blood at birth | 13 weeks
  The arterial umbilical cord blood concentration of glutathione will be measured in red blood cell lysates on C18-reverse phase column using liquid-chromatography combined to mass spectrometry. Homocysteine, cysteine, reduced (GSH) and oxidized (GSSG) glutathione levels will be measured in erythrocytes by comparing an experimental arm versus a placebo arm
Maternal blood concentrations of glutathione (micromoles/L) and their total antioxidant capacity at inclusion. | 18 weeks
  Changes in glutathione concentration (micromoles/L) in maternal red blood cells will be measured at inclusion and compared in an experimental arm versus a placebo arm. The maternal blood concentration of glutathione will be assessed as in the primary outcome measurement description. Total antioxidant capacity of maternal blood will be measured in plasma using kits such as Trolox Equivalent Antioxidant Capacity (TEAC) assay or lipid-peroxide secretion, measured by TBARS levels, combined to the measurement of levels of oxidized (carbonylated) proteins by mass spectrometry.
Maternal blood concentrations of glutathione (micromoles/L) and their total antioxidant capacity at delivery, following antenatal NAC supplementation. | 18 weeks
  Changes in glutathione concentration (micromoles/L) in maternal red blood cells will be measured at delivery and compared in an experimental arm versus a placebo arm. The maternal blood concentration of glutathione will be assessed as in the primary outcome measurement description. Total antioxidant capacity of maternal blood will be measured in plasma using kits such as Trolox Equivalent Antioxidant Capacity (TEAC) assay or lipid-peroxide secretion, measured by TBARS levels, combined to the measurement of levels of oxidized (carbonylated) proteins by mass spectrometry.
Placental total antioxidant capacity at delivery | at delivery
  Placental gene expression patterns of various enzymes involved in oxidative status such as superoxide dismutase, catalase and glutathione peroxidase and reductase will be measured in an experimental arm versus a placebo arm. Levels of free radical scavengers such as glutathione will be measured using liquid-chromatography combined to mass spectrometry. Placental total antioxidant capacity will be measured using TEAC or TBARS assays, combined to the measurement of levels of oxidized (carbonylated) proteins.
Breast milk sulphur amino acid pattern on day 7 of the postpartum period following NAC supplementation. | 19 weeks
  Colostrum or native breastmilk collected at day 7 will serve for determination of glutathione levels and other sulphur amino acids measured using liquid-chromatography combined to mass spectrometry.
Total antioxidant capacity on day 7 of the postpartum period following NAC supplementation. | 19 weeks
  Total antioxidant capacity will be measured using TEAC or TBARS assays in combination with mass spectrometry assessment of oxidized (carbonylated) proteins.
Maternal metabolome and lipidome at delivery following the antenatal NAC supplementation. | 18 weeks
  Metabolomic, lipidomic and amino acid patterns will be measured in maternal blood at GSH MAP-inclusion and at delivery using liquid-chromatography combined to mass spectrometry. The significance of the impact of NAC supplementation on these patterns will be assessed in link with maternal clinical data.
Weight variations | Hospital discharge (4 months)
  Weight will be evaluated in the fetus by maternal ultra-sound scans and measured on the newborn at birth and during his hospital stay. The significance of the impact of antenatal NAC supplementation on the anthropometric fetal and newborn data will be assessed taking into account clinical data.
Lenght variations | Hospital discharge (4 months)
  Length will be evaluated in the fetus by maternal ultra-sound scans and measured on the newborn at birth and during his hospital stay. The significance of the impact of antenatal NAC supplementation on the anthropometric fetal and newborn data will be assessed taking into account clinical data.
Head circumference variations | Hospital discharge (4 months)
  Head circumference will be evaluated in the fetus by maternal ultra-sound scans and measured on the newborn at birth and during his hospital stay. The significance of the impact of antenatal NAC supplementation on the anthropometric fetal and newborn data will be assessed taking into account clinical data.
Postnatal follow up of newborn blood concentration of glutathione during his first days of life. | from birth until hospital discharge (4 months)
  Newborn blood currently collected for clinical assessment during hospitalization will be analyzed in order to determine glutathione using liquid-chromatography combined to mass spectrometry. .
Postnatal follow up of newborn blood concentration of total antioxidant capacity during his first days of life. | from birth until hospital discharge (4 months)
  Newborn blood total antioxidant capacity will be measured using TEAC or TBARS assays.
Postnatal follow up of newborn blood concentration of and metabolome/lipidome during his first days of life. | from birth until hospital discharge (4 months)
  Newborn blood currently collected for clinical assessment during hospitalization will be analyzed in order to determine metabolome/lipidome using liquid-chromatography combined to mass spectrometry.
Improvement of the clinical outcome of the newborn until discharge from hospital. | 4 months
  Clinical data in newborn until his discharge and frequency of postnatal pathologies associated with prematurity.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Küster, Dr, Principal Investigator — Nantes University Hospital Nantes
Locations (1):
- Chu de Nantes, Nantes, France